CLINICAL TRIAL: NCT04368221
Title: Characterization of Fungal Infections in COVID-19 Infected and Mechanically Ventilated Patients in ICU
Acronym: MY-CO-VID
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC20_8885_MY_CO_VID
Record Dates: First submitted 2020-04-24; First posted 2020-04-29 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Covid-19
Keywords: Invasives mycoses; aspergillosis; pneumocystosis; mucormycosis
MeSH Terms: conditions — COVID-19; Aspergillosis; Pneumonia, Pneumocystis; Mucormycosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Characterization of fungal infections in COVID-19 infected and mechanically ventilated patients in ICU

DETAILED DESCRIPTION:
Currently, ICU patients with ARDS, whatever the etiology, are not systematically screened for the detection of respiratory fungal infections.

Here, the protocol will be in two steps:

First step

COVID-19 patients hospitalized in ICU for ARDS will benefit for a systematic screening with a fungal respiratory syndromic panel once or twice a week from entry to discharge from ICU, with minimum 3 samples when discharge occurs after 15 days::

* Sample: tracheal aspiration, bronchial aspiration, BAL
* Fungal respiratory panel: samples will be processed in each lab for culture without direct examination nor stained smears, and real-time PCR will be performed for Aspergillus, Pneumocystis jirovecii and mucormycetes
* Results will be given to ICU in order to optimize the management of the patient Second step

Complementary analysis will be performed in order to finalize the diagnostic and to differentiate between colonization and infection, with:

* Serum detection of galactomannan and serum Aspergillus PCR in case of positive respiratory sample for Aspergillus
* Serum/plasma beta-D-glucan detection in case of positive respiratory sample for Pneumocystis jirovecii
* Serum mucorales PCR in case of positive respiratory sample for mucorales This second step is possible in most of the labs, but when necessary a confirmation test can be externalized. A process of DNA transmission to a reference lab within each region will be implemented.

This second step will allow to classify infections as probable or proven according to international recommendations.

Case report form (CRF) A short but standardized CRF will be proposed to all centers in order to collect demographic data and the essential clinical and laboratory data during the survey.

ELIGIBILITY:
Inclusion criteria :

* ICU patients COVID-19 diagnosed by RT-PCR
* Intubated and mechanically ventilated patients
* Adult patients
* Patients (or legal representative) informed on the research without opposition

Non-inclusion criteria :

* Patients <18 years old
* People of full age who are the subject of a judicial safeguard,

Exclusion criteria:

* Patient, or legal representative opposing the pursuit of the research
* Patients under judicial protection will be excluded as soon as the investigator becomes aware of their status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients hospitalized in ICU for ARDS
Sampling Method: Non-Probability Sample
Enrollment: 576 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Opportunistic fungal co-infections. | at 12 months
  Prevalence of opportunistic fungal co-infections.

SECONDARY OUTCOMES:
Median time | at 12 months
  Determination of the median time between entry in ICU and beginning of ARDS and (i) colonization and (ii) probable/proven infection with Aspergillus, Pneumocystis jirovecii and mucormycetes
Time between diagnosis and targeted treatment | at ICU discharge, up to 1 month
  Evaluation of the time between diagnosis and targeted treatment
Preventive strategies | At 12 months
  Number of proposals for evaluation of preventive strategies if necessary, because of high incidence, in terms of chemoprophylaxis and/or environmental measures

CONTACTS AND LOCATIONS:
Locations (22):
- France (22):
  - CHU Angers, Angers
  - CHU de Brest, Brest
  - CHU de Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CHU Lille, Lille
  - CHU Lyon, Lyon
  - CHU Marseille, Marseille
  - CHU Nantes, Nantes
  - CHU de Nice, Nice
  - CHU Paris - Avicenne, Paris
  - CHU Paris - Bichat, Paris
  - CHU Paris - HEGP, Paris
  - CHU Paris - Mondor, Paris
  - CHU Paris - Tenon, Paris
  - Hôpital Lariboisière/ St Louis, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours

REFERENCES:
- [Derived] Gangneux JP, Dannaoui E, Fekkar A, Luyt CE, Botterel F, De Prost N, Tadie JM, Reizine F, Houze S, Timsit JF, Iriart X, Riu-Poulenc B, Sendid B, Nseir S, Persat F, Wallet F, Le Pape P, Canet E, Novara A, Manai M, Cateau E, Thille AW, Brun S, Cohen Y, Alanio A, Megarbane B, Cornet M, Terzi N, Lamhaut L, Sabourin E, Desoubeaux G, Ehrmann S, Hennequin C, Voiriot G, Nevez G, Aubron C, Letscher-Bru V, Meziani F, Blaize M, Mayaux J, Monsel A, Boquel F, Robert-Gangneux F, Le Tulzo Y, Seguin P, Guegan H, Autier B, Lesouhaitier M, Pelletier R, Belaz S, Bonnal C, Berry A, Leroy J, Francois N, Richard JC, Paulus S, Argaud L, Dupont D, Menotti J, Morio F, Soulie M, Schwebel C, Garnaud C, Guitard J, Le Gal S, Quinio D, Morcet J, Laviolle B, Zahar JR, Bougnoux ME. Fungal infections in mechanically ventilated patients with COVID-19 during the first wave: the French multicentre MYCOVID study. Lancet Respir Med. 2022 Feb;10(2):180-190. doi: 10.1016/S2213-2600(21)00442-2. Epub 2021 Nov 26. PMID 34843666